CLINICAL TRIAL: NCT05009797
Title: PROSPective Evaluation of Outcome After CatheTer Ablation in Atrial Fibrillation : LONGITUDINAL STUDY OF PATIENTS UNDERGOING RADIOFREQUENCY ABLATION OF ATRIAL FIBRILLATION.
Brief Title: PROSPective Evaluation of Outcome After CatheTer Ablation in Atrial Fibrillation
Acronym: PROSPECT-AF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_83; 2020-A02171-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Arrhythmia; Biomarkers
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat, plasma, serum, PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing atrial fibrillation catheter ablation: Patients undergoing scheduled atrial fibrillation catheter ablation.
  Interventions: Procedure: atrial fibrillation catheter ablation

INTERVENTIONS:
Procedure: atrial fibrillation catheter ablation — The ablation is performed under local anesthesia or general anesthesia. A transseptal puncture will be performed to access the left atrium. Pulmonary vein isolation will be performed as a first step. Additional lesions will be made at the discretion of the operators. Patients will receive anticoagulation for at least 3 months after the ablation. Treatment thereafter will be extended at the discretion of the treating physician.

SUMMARY:
Atrial fibrillation ablation is the most common intervention performed worldwide. Up to 20 to 45% of patients show recurrence of AF within 12 month after catheter ablation, however its determinant are incompletely understood.

The aim of the PROSPECT-AF study is to assess the predictors of AF recurrence within the 3 years following ablation using clinical variables and innovative biomarkers in a prospective cohort of 750 patients undergoing atrial fibrillation catheter ablation.

The secondary aims are to assess the incidence of major adverse cardiovascular outcomes (MACE) and the incidence of major bleeding within the 3 years Wolfing catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing atrial fibrillation catheter ablation
* Able to give their consent

Exclusion Criteria:

* Childs
* Patient under guardianship
* Patients unable to give their consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Lille University Hospital for schedulled Atrial fibrillation catheter ablation
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation recurrence. | At 3 years

SECONDARY OUTCOMES:
Incidence of major adverse cardiovascular events (MACE) including hospitalization for acute heart failure, cardiovascular death, stroke, myocardial infarction | At 3 years
Incidence of major bleeding (defined by BARC≥3 bleeding) | At 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Ninni, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Institut Coeur-Poumon, CHU, Lille, France